CLINICAL TRIAL: NCT06122896
Title: Prospective Screening for Pancreatic Ductal Adenocarcinoma in High-Risk Individuals
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Matthew B. Yurgelun, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-147
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma; Pancreatic Neoplasm
Keywords: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma; Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endosonography; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pancreatic Cancer High-Risk Participants (Experimental): Study procedures will be conducted as follows:
  * Baseline visit with questionnaires, blood tests, and pancreas screening procedure (EUS or MRI/MRCP).
  * Pancreas screening procedures (Endoscopic ultrasound (EUS), or Magnetic Resonance (MRI)/Magnetic Resonance Cholangiopancreatography (MRCP), and collection of blood, stool, and saliva samples) every 12 months.
  * Blood tests and questionnaires every 6 months.
  * Follow up visits.
  Interventions: Other: Screening Blood Tests; Diagnostic Test: Endoscopic Ultrasound; Combination Product: Magnetic Resonance Imaging; Combination Product: Magnetic Resonance Cholangiopancreatography

INTERVENTIONS:
Other: Screening Blood Tests — Carbohydrate antigen (CA) 19-9, and Hemoglobin A1C (HbA1c) per standard-of-care.
Diagnostic Test: Endoscopic Ultrasound — Annually and per National Comprehensive Cancer Network Guidelines (NCCN) guidelines.
  Other Names: EUS
Combination Product: Magnetic Resonance Imaging — Annually and per National Comprehensive Cancer Network Guidelines (NCCN) guidelines.
  Other Names: MRI
Combination Product: Magnetic Resonance Cholangiopancreatography — Annually and per National Comprehensive Cancer Network Guidelines (NCCN) guidelines.
  Other Names: MRCP

SUMMARY:
The purpose of this research is to see if adding blood-based tests and symptom review to standard-of-care pancreatic cancer screening procedures can identify cancer early among individuals with increased risk.

DETAILED DESCRIPTION:
In this research study, investigators will combine blood-based tests and review of symptoms with standard-of-care pancreatic cancer screening procedures to see if pancreatic cancer can be detected early among individuals with increased risk. Pancreatic cancer screening procedures include Endoscopic Ultrasound (EUS), Magnetic Resonance Imaging (MRI), or Magnetic Resonance Cholangiopancreatography (MRCP).

The research study procedures include screening for eligibility, questionnaires, clinic visits, endoscopic ultrasound (EUS) or Magnetic Resonance (MRI)/Magnetic Resonance Cholangiopancreatography (MRCP), and collection of blood, stool, and saliva samples.

Participation in this research study will be a minimum of 30 months and up to 20 years via review of medical records and the annual collection of blood and stool samples.

It is expected that about 5,000 people will take part in this research study.

This study is supported by the Hale Family Research Center at Dana-Farber Cancer Institute.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet any of the following:

* Individuals with pathogenic/likely pathogenic germline variants in STK11, and age ≥30 years.
* Individuals with pathogenic/likely pathogenic germline variants in CDKN2A, and age ≥40 years (or 10 years younger than the earliest exocrine pancreatic cancer diagnosis in the family, whichever is earlier).
* Individuals with pathogenic/likely pathogenic germline variants in one of the other pancreatic cancer susceptibility genes (ATM, BRCA1, BRCA2, MLH1, MSH2, MSH6, EPCAM, PALB2, TP53), and age ≥50 years (or 10 years younger than the earliest exocrine pancreatic cancer diagnosis in the family, whichever is earlier) AND

  • Exocrine pancreatic cancer in ≥1 first- or second-degree relative from the same side of (or presumed to be from the same side of) the family as the identified pathogenic/likely pathogenic germline variant.
* Individuals with pathogenic/likely pathogenic variants in PRSS1 AND a clinical phenotype consistent with hereditary pancreatitis, and age ≥40 years (or 20 years after onset of pancreatitis, whichever is earlier).
* Individuals with familial pancreatic cancer including:

  * Family history of exocrine pancreatic cancer in ≥2 first-degree relatives from the same side of the family, even in the absence of a known pathogenic/likely pathogenic germline variant, OR
  * Family history of exocrine pancreatic cancer in 1 affected first-degree relative and 1 second-degree relative, even in the absence of a known pathogenic/likely pathogenic germline variant, OR
  * Family history of exocrine pancreatic cancer in ≥3 first- and/or second-degree relatives from the same side of the family, even in the absence of a known pathogenic/likely pathogenic germline variant.
* Individuals who are undergoing clinically recommended pancreatic cancer surveillance.

Exclusion Criteria:

* Individuals with active or prior pancreatic ductal adenocarcinoma diagnosis.
* Individuals with any active metastatic cancer.
* Individuals who are unable to give informed consent.
* Individuals who are under the age of 18 (infants, children, teenagers).
* Individuals unable to tolerate Magnetic Resonance Imaging/Magnetic Resonance Cholangiopancreatography and Endoscopic Ultrasound.
* Pregnant women are unlikely to be undergoing screening procedures and will not be considered eligible but can consent to the study at a later date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2040-10-31 (Estimated); Study Completion 2041-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Incident Pancreatic Cancers or High-Grade Pancreatic Neoplasms | 6-monthly for 3 years with 5-year follow-up
  Subjects will be counted in this metric if they have pathological tissue confirmation of a pancreatic cancer or high-grade dysplasia during each observation period.
Number of Imaging-Positive Pancreatic Cancers or High-Grade Neoplasms | 6-monthly for 3 years with 5-year follow-up
  Subjects will be considered imaging-positive if they have a biopsy-confirmed pancreatic ductal adenocarcinoma or high-grade dysplasia that was initially detected on standard-of-care screening MRI or EUS during each observation period.
Number of Imaging-Negative, Assay-Positive Pancreatic Cancers or High-Grade Neoplasms | 6-monthly for 3 years with 5-year follow-up
  Subjects will be considered imaging-negative and assay-positive if: 1) the subject has a study visit that yields any newly positive CA19-9 (>35U/mL or >=20% increase) or diabetes (FBG >100mg/dL for first time or HgbA1c increased by 0.5) assay result or ENDPAC score >=3 with negative MRI and/or EUS at that visit or within six months prior to that visit; and 2) has a biopsy-confirmed pancreatic ductal adenocarcinoma or high-grade dysplasia within two years after that visit.

SECONDARY OUTCOMES:
Positive Predictive Value of Blood Assays | 6-monthly for 3 years
  Positive predictive value of blood assays, defined as newly positive CA19-9 (>35U/mL or >=20% increase) or diabetes (FBG >100mg/dL for first time or HgbA1c increased by 0.5) assay result or ENDPAC score >=3, with a positive biopsy for PDAC or High-Grade Dysplasia within six months divided by the total number with a positive blood assay.
Negative Predictive Value of Blood Assays | 6-monthly for 3 years
  Negative predictive value of blood assays, defined as CA19-9 (<=35U/mL or <20% increase) or diabetes (FBG <100mg/dL for first time or HgbA1c increased by less than 0.5) assay result or ENDPAC score <3, without a positive biopsy for PDAC or High-Grade Dysplasia within six months divided by the total number with a negative blood assay.
Proportion of Screen-Detected, Resected Pancreatic Lesions | 6-monthly for 3 years
  Number of screen-detected pancreatic lesions that are resected compared to the total number of screen-detected pancreatic lesions.
Proportion of Non-Worrisome Pancreatic Lesions | 6-monthly for 3 years
  Number of pancreatic lesions that are biopsied without cancer or high-grade dysplasia divided by number of pancreatic lesions that are biopsied.
Incremental Yield of Blood-Based Assays over Standard-of-Care Screening | 6-monthly for 3 years
  Number of imaging-negative, assay-positive cases showing cancer or high-grade dysplasia divided by the total number of imaging-negative cases with cancer or high-grade dysplasia.
Number of False-Positive Assay Results | 6-monthly for 3 years
  Number of positive assay results, defined as newly positive CA19-9 (>35U/mL or >=20% increase) or diabetes (FBG >100mg/dL for first time or HgbA1c increased by 0.5) assay result or ENDPAC score >=3, without a clinical diagnosis of pancreatic cancer within one year.
Number of Non-PDAC Cancer Diagnoses | 6-monthly for 3 years
  Number of non-PDAC cancer detected through blood-based assays, EUS and/or MRI during the active screening period.
Clinical Predictors of Neoplastic Development | up to 8 years
  Frequencies of clinical predictors of neoplastic development as indicated by responses to the study surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Yurgelun, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Matthew Yurgelun, Matthew_Yurgelun@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu